CLINICAL TRIAL: NCT04512014
Title: Evaluation of Lactate Levels in as a Risk Factor for Posthepatectomy Liver Failure
Brief Title: Perioperative Lactate Kinetics in Patient Undergoing Major Liver Surgery
Status: Completed | Type: Observational
Sponsor: Institutul Clinic Fundeni (Other)
Responsible Party: Principal Investigator, Popescu Mihai, Clinical Professor, Institutul Clinic Fundeni
Other Study IDs: Liver_lactate
Record Dates: First submitted 2020-08-10; First posted 2020-08-13 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Liver Failure, Acute
MeSH Terms: conditions — Liver Failure, Acute

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- major liver surgery: Patients undergoing major liver surgery
  Interventions: Diagnostic Test: serum lactate

INTERVENTIONS:
Diagnostic Test: serum lactate — perioperative measurement of lactate levels

SUMMARY:
Major liver surgery is associated with increased incidence of perioperative complications and increased mortality if these are not addressed quickly in a high dependency intensive care unit. Of these, posthepatectomy liver failure (PHLF) represents one of the most important cause of postoperative unfavourable outcome. The present study investigates the correlation between lactate levels and PHLF. Lactate levels were collected at six specific timepoints: preoperative, pre-dissection phase, post-dissection phase, end of surgery and 24-hours and 48-hours in the postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing major liver surgery for primary or secondary tumours

Exclusion Criteria:

* unsigned patient consent
* death within 24 hours
* need for perioperative renal replacement therapy
* underlying liver disease (e.g. liver cirrhosis)
* other causes of raised lactate levels (e.g. shock)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients undergoing major liver failure in our institution
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
lactate levels (mmol/L) in patients with PHLF | early postoperative period (48 hours)
  correlation of lactate levels with the diagnosis of PHLF

SECONDARY OUTCOMES:
mortality | 30 days mortality
  in hospital mortality

CONTACTS AND LOCATIONS:
Overall Officials: Dana Tomescu, Prof, Study Chair — Fundeni Clinical Institute
Locations (1):
- Fundeni Clinical Institute, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: No